CLINICAL TRIAL: NCT06745427
Title: A Multi-center Prospective Study on the Oncological and Reproductive Outcomes and Quality of Life in Young Woman After Fertility-sparing Treatment of Endometrial Cancer and Endometrial Intraepithelial Hyperplasia
Acronym: PreFerEC/EIN
Status: Not yet recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Charlotta Riese, MD, Region Stockholm
Other Study IDs: 2024048701
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Endometrial Cancer; Endometrial Intraepithelial Neoplasia; Fertility-sparing Surgery
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We will investigate the safety and efficiency of fertility-sapring treatment in ypung women witg endometrial cancer and endometrial intraepithelial hyperplasia

DETAILED DESCRIPTION:
A multi-center prospective study on the oncological and reproductive outcomes and quality of life in young woman after fertility-sparing treatment of endometrial cancer and endometrial intraepithelial hyperplasia

ELIGIBILITY:
Inclusion Criteria:

* Fertility sparing treatment of EC and EIN.
* 18-45 Years old
* From start study (Jan 2025 - end study Jan 2028)
* All centras in Sweden

Exclusion Criteria:

* Not English och Swedish speaking

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2028-01-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Relaps of endometrial cancer or EIN after fertility-sparing treatment | from enrollment to 2 years after fertility-sparing treatment
  Relaps of endometrial cancer or EIN after fertility-sparing treatment

SECONDARY OUTCOMES:
Live birth rate in women that has been treated with fertility-sparing treatment for EC or EIN | From start of study to 2 years after fertility-sparing treatment
  Live birth rate in women that has been treated with fertility-sparing treatment for EC or EIN

IPD SHARING:
Plan to Share IPD: Undecided